CLINICAL TRIAL: NCT05579574
Title: An Open-Label, Single-Sequence, Crossover Study to Investigate the Interaction of Multiple Doses of BMS-986322 at Steady State and Multiple Doses of a Combined Oral Hormonal Contraceptive (Ethinyl Estradiol/Norethindrone) in Healthy Female Participants
Brief Title: A Study to Investigate the Interaction of BMS-986322 and a Combined Oral Hormonal Contraceptive (Ethinyl Estradiol [EE]/Norethindrone [NET]) in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM032-030
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Healthy Participants
Keywords: BMS-986322; Loestrin; Combined oral hormonal contraceptive; Ethinyl Estradiol; Norethindrone; Drug-drug interaction
MeSH Terms: interventions — norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986322 and Loestrin (Experimental): Loestrin, then progress to combination
  Interventions: Drug: BMS-986322; Drug: Loestrin

INTERVENTIONS:
Drug: BMS-986322 — Specified dose on specified days
Drug: Loestrin — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the effect of multiple doses of BMS-986322 on the pharmacokinetics (PK) of Loestrin components in healthy female participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, defined as having no clinically significant active or ongoing medical condition, physical examination abnormality, abnormal ECG finding, and abnormal clinical laboratory determinations that in the opinion of the investigator would compromise the conduct, results, or interpretation of the study findings.
* Have a negative QuantiFERON®-TB Gold test result at screening or documentation of a negative result within 4 weeks prior to the start of study intervention.
* Have a normal renal function at screening as evidenced by an estimated glomerular filtration rate (eGFR) ≥ 80 milliliter (mL)/minute (min)/1.732m^2 calculated with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Any acute infection or febrile illness within 7 days before Day 1 of Cycle 2.
* Any history or risk for tuberculosis (TB), specifically participants with 1) current clinical, radiographic or laboratory evidence of active TB; 2) history of active TB unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; latent TB that has not been successfully treated.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for EE/NET | Up to 28 days
Cmax for EE/NET with BMS-986322 | Up to 28 days
Area under the concentration-time curve in 1 dosing interval (AUC[tau]) for EE/NET | Up to 28 days
AUC (tau) for EE/NET with BMS-986322 | Up to 28 days

SECONDARY OUTCOMES:
Cmax for BMS-986322 | Up to 31 days
Cmax for BMS-986322 with EE/NET | Up to 31 days
AUC (tau) for BMS-986322 | Up to 31 days
AUC (tau) for BMS-986322 with EE/NET | Up to 31 days
Number of participants with Adverse Events (AEs) | Up to 119 days
Number of participants with Serious AEs (SAEs) | Up to 119 days
Number of participants with physical examination abnormalities | Up to 119 days
Number of participants with vital sign abnormalities | Up to 119 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 119 days
Number of participants with clinical laboratory abnormalities | Up to 119 days
Time of maximum observed plasma concentration (Tmax) for EE/NET | Up to 28 days
Tmax for EE/NET with BMS-986322 | Up to 28 days
Tmax for BMS-986322 | Up to 31 days
Tmax for BMS-986322 with EE/NET | Up to 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 0001, Anaheim, California
  - Local Institution - 0002, Anaheim, California

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com